CLINICAL TRIAL: NCT07227025
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of Amivantamab and Olomorasib Combination Therapy in Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Amivantamab and Olomorasib Combination Therapy in Participants With Metastatic Non-Small Cell Lung Cancer
Acronym: KaRAnaSa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 61186372PANSC2004; 61186372PANSC2004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase 1: Combination Dose Selection (Experimental): Participants will receive amivantamab along with olomorasib to determine the RP2CD of the combination therapy until disease progression, significant toxicity, or until another criterion for discontinuation of study treatment is met. Eligible participants may have the option to transfer to a long-term extension (LTE) phase for continued access to study treatments.
  Interventions: Drug: Amivantamab; Drug: Olomorasib
- Phase 2: Expansion (Experimental): Participants will receive amivantamab and olomorasib combination therapy at the RP2CD determined in Phase 1 until disease progression, significant toxicity, or until another criterion for discontinuation of study treatment is met. Eligible participants may have the option to transfer to LTE phase for continued access to study treatments.
  Interventions: Drug: Amivantamab; Drug: Olomorasib

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered.
  Other Names: JNJ-61186372; RYBREVANT
Drug: Olomorasib — Olomorasib will be administered.
  Other Names: LY3537982

SUMMARY:
The main purpose of this study is to find out the most suitable dose (recommended phase 2 combination dose [RP2CD]) of amivantamab and olomorasib combination therapy and to assess how well the combination slows down or prevents the growth of tumors in participants with KRAS G12C mutant metastatic non-small cell lung cancer (NSCLC: the most common type of lung cancer; metastatic: has spread to other parts of the body; KRAS G12C mutant: mutation [change] in the kirsten rat sarcoma viral oncogene homolog [KRAS] gene in tumor cells in which glycine [G] at position 12 is replaced with cystine [C]).

ELIGIBILITY:
Inclusion criteria:

* Participant must have histologically or cytologically confirmed metastatic NSCLC characterized by a KRAS G12C mutation at the time of enrollment. For Phase 1: Participant must have progressed on or after, or have intolerance to, platinum-based chemotherapy and Programmed Death-Ligand 1 (PD-L1)-targeted immunotherapy given in combination or sequentially. Receipt of additional lines of prior therapy is permitted. Progression must have occurred on or after the most recent line of systemic anticancer therapy. For Phase 2: Participant must have progressed on or after platinum-based chemotherapy and PD-L1-targeted immunotherapy given in combination or sequentially. Progression must have occurred on or after the most recent line of systemic anticancer therapy. Receipt of additional lines of prior therapy is not permitted
* Participant must have at least 1 measurable lesion, according to RECIST version.1.1, that has not been previously irradiated
* May have brain metastases only if previously definitively, locally treated, and participant is clinically stable and asymptomatic for greater than (>) 2 weeks and is off or receiving low-dose corticosteroid treatment for at least 2 weeks prior to start of study treatment
* Can have a prior or concurrent second malignancy (other than the disease under study) with natural history or treatment course that is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion criteria:

* Participant has history of uncontrolled illness
* Suspected or known allergies, hypersensitivity, or intolerance to amivantamab excipients or olomorasib excipients
* Medical history of (non-infectious) interstitial lung disease (ILD)/pneumonitis, or has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Presence of primary driver mutations (epidermal growth factor receptor [EGFR], anaplastic lymphoma kinase [ALK], mesenchymal-epithelial transition [MET], human epidermal growth factor receptor 2 [HER2], ROS1, neurotrophic tyrosine receptor kinase [NTRK], B-Raf proto-oncogene [BRAF], rearranged during Transfection [RET], neuroblastoma RAS viral oncogene homolog [NRAS], and other KRAS mutations besides G12C) as determined by local genomic testing
* Prior treatment with any KRAS inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse Events (AEs) by Severity | Up to approximately 3 years 2 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An assessment of severity grade will be made by the investigator according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 defined as follows: Grade 1 (mild; asymptomatic or mild symptoms; intervention not indicated); Grade 2 (moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living [ADL]); Grade 3 (severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 (life-threatening consequences; urgent intervention indicated); Grade 5 (Death related to adverse event).
Phase 1: Number of Participants with Dose-Limiting Toxicities (DLTs) | Up to approximately 3 years 2 months
  DLT is defined as drug related adverse events and includes unacceptable non-hematologic toxicity, hematologic toxicity, pulmonary toxicity, or elevations in hepatic enzymes suggestive of drug-induced liver injury of Grade 3 or higher. Toxicities will be graded for severity according to the NCI-CTCAE, version 5.0.
Phase 2: Confirmed Objective Response Rate (ORR) | Up to approximately 3 years 2 months
  ORR is defined as the percentage of participants who achieve either a confirmed partial response (PR) or complete response (CR), using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 by investigator review. Confirmatory analysis may be performed using Blinded Independent Central Review (BICR).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) by Severity | Up to approximately 3 years 2 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An assessment of severity grade will be made by the investigator according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 defined as follows: Grade 1 (mild; asymptomatic or mild symptoms; intervention not indicated); Grade 2 (moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living [ADL]); Grade 3 (severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 (life-threatening consequences; urgent intervention indicated); Grade 5 (Death related to adverse event).
Number of Participants with Abnormalities in Clinical Laboratory Parameters | Up to approximately 3 years 2 months
  Number of participants with abnormalities in clinical laboratory values (which includes serum chemistry, hematology, coagulation, urinalysis, and serology) will be reported.
Phase 2: Duration of Response (DoR) | Up to approximately 3 years 2 months
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death from any case, whichever comes first, for participant who have PR or CR according to RECIST v1.1 by investigator review.
Phase 2: Disease Control Rate (DCR) | Up to approximately 3 years 2 months
  DCR is defined as the percentage of participants who achieve a PR, CR, or stable disease using RECIST v1.1.
Phase 2: Progression-Free Survival (PFS) | Up to approximately 3 years 2 months
  PFS is defined as the time from first dose date until the date of disease progression or death, whichever comes first, based on investigator assessment using RECIST v1.1 by investigator review.
Phase 2: Overall Survival (OS) | Up to approximately 3 years 2 months
  OS is defined as the time from the date of administration of the first dose of study treatment until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- United States (2):
  - New York University Langone Medical Center, New York, New York
  - Virginia Cancer Specialists, Fairfax, Virginia
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Shanghai East Hospital, Shanghai, China
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency